CLINICAL TRIAL: NCT01119833
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Pharmacokinetics of GMI-1070, A Pan-Selectin Inhibitor, In Subjects Hospitalized For Sickle Cell Vaso-Occlusive Crisis
Brief Title: Study of GMI-1070 for the Treatment of Sickle Cell Pain Crisis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GMI-1070-201
Record Dates: First submitted 2010-05-05; First posted 2010-05-10 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Crisis; Pain Crisis
Keywords: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — rivipansel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GMI-1070 (Experimental)
  Interventions: Drug: GMI-1070
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GMI-1070 — Intravenous GMI-1070 given twice a day during hospital stay for sickle cell pain crisis
  Arms: GMI-1070
Drug: Placebo — Intravenous Placebo given twice a day during hospital stay for sickle cell pain crisis
  Other Names: saline placebo
  Arms: Placebo

SUMMARY:
GMI-1070 is a new drug that may reduce the stickiness of cells in the blood. The purpose of this study is to evaluate whether GMI-1070 can reduce the time it takes for pain to go away in patients with vaso-occlusive crisis (also known as a sickle cell pain crisis). The study will also collect information on the safety of GMI-1070, how much of the drug is in the blood and urine, and if there are any other effects when used in patients who are in the hospital for a sickle cell pain crisis.

DETAILED DESCRIPTION:
Patients being admitted to the hospital for pain crisis may be eligible for this study. In addition, patients should be 12-60 years old and have sickle cell types SS or S-beta-thalassemia. People who take part in the study will be evaluated and then randomly assigned to receive either GMI-1070 or a placebo by IV, in addition to all other usual treatments for their pain crisis.

During the hospital stay for pain crisis, GMI-1070 or placebo will be given twice a day, and patients will be asked about their pain severity (pain score) at the beginning of the study and every few hours during their hospital stay. Their general health, vital signs, lab tests, and pain medications will also be checked on a regular basis through the hospital stay. When a patient is feeling well enough to go home, the study drug (GMI-1070 or placebo) will be stopped, and the patient may go home. Participants will be asked to come back to clinic for a check-up a few days after leaving the hospital, and one month after leaving the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. 12 to 60 years of age
2. Confirmed diagnosis of sickle cell disease (HbSS or HbS-β0thalassemia)
3. Diagnosis of VOC at the time of enrollment
4. Hospitalized or in process of admission at the time of enrollment
5. Able to receive the first dose of study drug within 24 hours of initial medical evaluation in the Emergency Department/clinic for VOC;

   o Subjects treated as an outpatient within the past 48 hours for the same VOC episode may be enrolled if dosing is also expected within 24 hours of their second (admitting) presentation.
6. Documented and observed written informed consent (and assent, where applicable)

Exclusion Criteria:

1. Infection, diagnosed or strongly suspected, as evidenced by one or more of the following:

   * Fever >39°C (102.2°F)
   * In the presence of fever ≥38.5°C (101.3°F), 1 of the following:

     * Positive findings (suspicious for infection) on diagnostic tests, such as cerebral spinal fluid [CSF] evaluation, radiographs, or bacterial culture of normally sterile sites
     * Exam findings leading to diagnosed or strongly suspected bone or joint infection
     * Determination by physician that bacterial or serious systemic viral infection is likely (eg, influenza, mononucleosis)
     * Subjects may be included with uncomplicated urinary tract infections (provided they do not have fever ≥38.5° C [101.3° F] or costo-vertebral angle [CVA] tenderness), and/or suspected minor viral syndromes (upper respiratory infection symptoms but no symptoms suggestive of bacterial infection other than uncomplicated otitis media or uncomplicated streptococcal pharyngitis)
2. Acute chest syndrome, diagnosed or strongly suspected, as evidenced by a new infiltrate on chest radiograph, and 1 or more of the following:

   * Fever >39° C (102.2° F)
   * Hypoxia (confirmed by arterial blood gases [ABG] with paO2 <70 mmHg)
   * Chest pain
   * Suspicious findings on exam (tachypnea, intercostal retractions, wheezing, and/or rales)
3. Sickle cell disease (SCD) pain atypical of VOC, including hepatic or splenic sequestration, cholecystitis, or pneumonia.
4. Acute stroke, acute priapism, severe avascular necrosis of the hip/shoulder when the presenting pain is only in the affected hip/shoulder
5. Serum creatinine:

   * >1.2 mg/dL for subjects 16 to 60 years of age
   * >1.0 mg/dL for subjects 12 to 15 years of age
6. Alanine transaminase (ALT/SGPT) >2x upper limit of normal (ULN) (based on clinic laboratory normal range)
7. Hemoglobin <5 g/dL
8. Platelets <100,000/mm3
9. Recent (within the past 30 days) major surgery, hospitalization for other than VOC, documented serious bacterial infection requiring antibiotic treatment, or significant bleeding
10. Hospitalization for uncomplicated VOC, or treated with parenteral pain medications in other medical settings such as the emergency department or day hospital for uncomplicated VOC, within past 14 days.

    o Subjects may be included if treated as an outpatient within the past 48 hours for the same VOC episode.
11. Recent (within the past 90 days) cerebrovascular accident, transient ischemic attack, or seizure
12. pRBC transfusions in the past 14 days
13. Systemic steroid therapy within 48 hours prior to enrollment or expectation that therapy may be used during the study (inhaled or topical steroids are allowed)
14. For those on chronic or long-acting opioids, a change in dose in the past 14 days OR pain requiring medical attention in the past 14 days (change in opioid medication for acute pain in the past 48 hours and directly related to this VOC admission is allowed)
15. Greater than 5 episodes of hospitalization for VOC in the past 6 months (180 days)
16. Medical or psychiatric condition that, in the opinion of the investigator, may pose a risk to the subject for participation or interfere with the conduct or results of the study
17. Currently receiving, or has received within the previous 4 weeks, any other investigational agent
18. Previous administration of GMI-1070
19. Expectation that the subject will not be able to be followed for the duration of the study
20. Pregnant or lactating female; or female of childbearing potential or male unable or unwilling to comply with birth control methods or abstinence during the course of the study
21. Active use of illicit drugs and/or alcohol dependence, as determined by the investigator

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Reduction in time to resolution of vaso-occlusive crisis | Up to 7 days or resolution
  Including pain score, feeling ready to leave the hospital, and actual time of leaving the hospital

SECONDARY OUTCOMES:
Safety during the study | Up to 28 days post last dose
  Including changes in physical exam, lab tests, and vital signs
Pharmacokinetics | Baseline thru 36 hrs post last dose
  Pharmacokinetics including half-life and concentration of GMI-1070 in the blood and urine
Markers of inflammation and cell stickiness in the blood | Up thru 28 days post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn J Telen, MD, Principal Investigator — Duke University; Helen Thackray, MD, Study Director — GlycoMimetics, Inc.
Locations (22):
- United States (21):
  - University of Alabama Hospital, Birmingham, Alabama
  - Alta Bates Summit Medical Center, Berkeley, California
  - University of California, Davis Medical Center, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine, Miami, Florida
  - Georgia Health Sciences University, Augusta, Georgia
  - University of Illinois, Chicago, Chicago, Illinois
  - The Johns Hopkins School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - New York Methodist Hospital, Brooklyn, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Childrens' Hospital, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Rebelo AL, Chevalier MT, Russo L, Pandit A. Role and therapeutic implications of protein glycosylation in neuroinflammation. Trends Mol Med. 2022 Apr;28(4):270-289. doi: 10.1016/j.molmed.2022.01.004. Epub 2022 Feb 1. PMID 35120836
- [Derived] Telen MJ, Wun T, McCavit TL, De Castro LM, Krishnamurti L, Lanzkron S, Hsu LL, Smith WR, Rhee S, Magnani JL, Thackray H. Randomized phase 2 study of GMI-1070 in SCD: reduction in time to resolution of vaso-occlusive events and decreased opioid use. Blood. 2015 Apr 23;125(17):2656-64. doi: 10.1182/blood-2014-06-583351. Epub 2015 Mar 2. PMID 25733584
- [Derived] Deal watch: Pfizer deal for selectin inhibitor highlights potential of glycomimetic drugs. Nat Rev Drug Discov. 2011 Dec 1;10(12):890. doi: 10.1038/nrd3622. No abstract available. PMID 22129980